CLINICAL TRIAL: NCT05757388
Title: The Efficacy of Intraoperative Parecoxib Combined With Paracetamol for Reducing Opioid Consumption in Patients Undergoing Breast Cancer Surgery Under General Anesthesia: A Prospective Randomized Controlled Trial
Brief Title: Efficacy of Parecoxib Combined With Paracetamol in Mastectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HE641269
Record Dates: First submitted 2023-02-22; First posted 2023-03-07 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Post Operative Pain
Keywords: postoperative pain; multimodal anagesia
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib; Acetaminophen; Saline Solution

STUDY DESIGN:
Intervention Model Description: Group P receives the parecoxib 40 mg iv slowly push plus paracetamol 1 gm (100 mL) infusion drip in 30 min after induction or group C receives the normal saline in the same process.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Normal saline is prepared in the same packages as parecoxib and paracetamol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): Receives the parecoxib 40 mg iv slowly push plus paracetamol 1 gm (100 mL) infusion drip in 30 min after induction.
  Interventions: Drug: Parecoxib + paracetamol
- Group C (Placebo Comparator): Receives normal saline in the same process.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Parecoxib + paracetamol — Administers after induction of anesthesia.
  Other Names: Study drugs
  Arms: Group P
Drug: Normal saline — Administers after induction of anesthesia.
  Other Names: placebo
  Arms: Group C

SUMMARY:
Patients undergoing breast cancer surgery experience persistent pain after surgery and subsequent development of chronic pain. Parecoxib or paracetamol has been reported to reduce postoperative pain in mastectomy. The investigators aim to assess the effectiveness of the perioperative administration of parecoxib combined with paracetamol to reduce postoperative acute and subacute breast surgical pain.

DETAILED DESCRIPTION:
Patients with breast cancer undergoing mastectomy experience moderate postoperative pain which may persist for more than 3 months and may turn into chronic pain. This may interfere with the daily life of the patients. Proper prophylaxis and management to control postoperative pain are essential. Morphine is the most common drug to control postoperative pain. However, there are many serious side effects, e.g., nausea/vomiting, pruritus, ileus, constipation, sedation, and respiratory depression. Multimodal analgesia comprises the use of a combination of drugs to provide the opioid-sparing effect. Parecoxib, a selective cox-2 inhibitor, and intravenous paracetamol are reported to provide good postoperative analgesia. The investigators aim to apply a combination of parecoxib and paracetamol perioperatively to reduce postoperative morphine consumption.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer undergoing elective mastectomy
* ASA physical status 1-3

Exclusion Criteria:

* Allergy to parecoxib, paracetamol, or sulfonamide
* History of opioid use
* Pregnant
* Renal or hepatic disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine consumption | Up to 24 hours postoperatively
  Postoperative morphine requirement

SECONDARY OUTCOMES:
Postoperative pain score | Up to 3 months postoperatively
  Postoperative numeric rating score (0-10; higher score means a worse outcome) at rest and at movement
Postoperative nausea/vomiting score | Up to 24 hours postoperatively
  Postoperative nausea/vomiting score (0-3; higher score means a worse score)
Quality of life score | Up to 24 hours postoperatively
  WHOQOL-BREF-THAI questionair (World Health Organization Quality of Life Brief - Thai: 26-130; higher score means a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, MD, Study Chair — Khon Kaen University
Locations (1):
- Dr. Sirirat Tribuddharat, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Woolf CJ, Max MB. Mechanism-based pain diagnosis: issues for analgesic drug development. Anesthesiology. 2001 Jul;95(1):241-9. doi: 10.1097/00000542-200107000-00034. No abstract available. PMID 11465563
- [Background] Schug SA. The role of COX-2 inhibitors in the treatment of postoperative pain. J Cardiovasc Pharmacol. 2006;47 Suppl 1:S82-6. doi: 10.1097/00005344-200605001-00015. PMID 16785836
- [Background] Brett CN, Barnett SG, Pearson J. Postoperative plasma paracetamol levels following oral or intravenous paracetamol administration: a double-blind randomised controlled trial. Anaesth Intensive Care. 2012 Jan;40(1):166-71. doi: 10.1177/0310057X1204000121. PMID 22313079
- [Background] Nonaka T, Hara M, Miyamoto C, Sugita M, Yamamoto T. Comparison of the analgesic effect of intravenous acetaminophen with that of flurbiprofen axetil on post-breast surgery pain: a randomized controlled trial. J Anesth. 2016 Jun;30(3):405-9. doi: 10.1007/s00540-016-2150-0. Epub 2016 Feb 16. PMID 26882922
- [Background] Schug SA, Parsons B, Li C, Xia F. The safety profile of parecoxib for the treatment of postoperative pain: a pooled analysis of 28 randomized, double-blind, placebo-controlled clinical trials and a review of over 10 years of postauthorization data. J Pain Res. 2017 Oct 10;10:2451-2459. doi: 10.2147/JPR.S136052. eCollection 2017. PMID 29066931